CLINICAL TRIAL: NCT05497661
Title: Ultrasound Patellar Tendon Assessment and Thermography After 448kilohertz Capacitive Resistive Radiofrequency Stimulation in a Sporty Population
Brief Title: Ultrasound Patellar Tendon Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María Aguilar García, Principal Investigator, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UGranadaPatellarTendon
Record Dates: First submitted 2022-07-10; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Patellofemoral Pain; Ultrasonography
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of Capacitive Resistive Monopolar Radiofrequency in patellar tendon (Experimental): 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the dominant patellar tendon.
  Interventions: Other: 448kilohertz Capacitive Resistive Radiofrequency Stimulation in a Sporty Population.; Other: Placebo comparator
- Placebo Comparator: Placebo Monopolar Radiofrequency stimulus (Placebo Comparator): To simulate the application of Monopolar Radiofrequency stimulus on the dominant patellar tendon
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: 448kilohertz Capacitive Resistive Radiofrequency Stimulation in a Sporty Population. — 448kilohertz Capacitive Resistive Radiofrequency Stimulation on Patellar tendon in a Sporty Population.
  Arms: Effects of Capacitive Resistive Monopolar Radiofrequency in patellar tendon
Other: Placebo comparator — To simulate a 448kilohertz capacitive resistive monopolar radiofrequency application on the non dominant patellar tendon

SUMMARY:
448kilohertz capacitive resistive monopolar radiofrequency is a novel technique in physiotherapy and its usefulness and clinical relevance is still to be investigated at both clinical practice and also in performance. Current studies show promising results in different musculoskeletal disorders, however there no studies in the assessment of quality soft tissue in sporty population after the used of this technique.

DETAILED DESCRIPTION:
Patellar tendon injuries is is one of the most common musculoskeletal disorders, presenting a high prevalence in sport populations. Many factors have been proposed as the cause of pain and dysfunction, however there are no studies analysing possibilities of preventing patellar tendon injuries by using a radiofrequency stimulus.

The use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment looking for improve the quality of the tissue is still to be explored.

The hypothesis of the present project is that focus treatments on 448kilohertz capacitive resistive monopolar radiofrequency on the patellar tendon will produce better outcomes in terms of ultrasound assessment measured by quantified elastography, and this will decreased the possibilities of get injured.

The stimulus will be carried out on the patellar tendon region. All interventions will be developed by the same examiner, who is a physiotherapist with 6 years of clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Sporty people with at least 3 days of training per week

Exclusion Criteria:

* Suffer from knee pain.
* Sedentary people

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10-14 (Estimated); Primary Completion 2023-06-14 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in patellar tendon measured by quantified elastography imaging at 3 months [ Time Frame: Time Frame: time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)] ] | Time Frame: time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  The elastography is obtained when the anatomic image on grayscale ultrasound overlaps parametric color image that expresses the rate of deformity of the tissues, soft tissues tend to develop greater deformity and tissue deformity have lower rigidity

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Navarro Ledesma, Principal Investigator — University of Malaga; Ana González Muñoz, Study Chair — University of Malaga
Locations (1):
- Clínica Ana González, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No